CLINICAL TRIAL: NCT06773026
Title: A Phase 2, Open-label, Fixed-dose Study to Assess the Efficacy of Sodium Phenylbutyrate (ACER-001) in Treating Pediatric and Adult Patients With Medium Chain Acyl-CoA Dehydrogenase (MCAD) Deficiency Resulting From the Prevalent ACADM c.985 A>G (K304E) Mutation
Brief Title: Study of Sodium Phenylbutyrate (ACER-001) for the Treatment of Pediatric and Adults Patients With Medium Chain Acyl-CoA Dehydrogenase Deficiency (MCADD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jerry Vockley, MD, PhD (Other)
Collaborators: Zevra Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Jerry Vockley, MD, PhD, Chief, Division of Genetic and Genomic Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24100064
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Medium-chain Acyl-CoA Dehydrogenase Deficiency
Keywords: Medium-chain Acyl-CoA Dehydrogenase Deficiency
MeSH Terms: conditions — Medium chain acyl CoA dehydrogenase deficiency | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 4.0 g/m2/day BID sodium phenylbutyrate (Experimental): Up to 24 subjects (12: ages 4-9 years old; 12:10 years of age and older) will be randomized to take 4.0 g/m2/day divided into two daily doses
  Interventions: Drug: Sodium phenylbutyrate

INTERVENTIONS:
Drug: Sodium phenylbutyrate — Open-label design with doses of sodium phenylbutyrate at 4.0 g/m2/day
  Other Names: Olpruva

SUMMARY:
This is a medical research study to test a medication in patients 4 years of age and older with a disease called medium-chain acyl-CoA dehydrogenase deficiency (MCADD) caused by the common ACADM c.985 A>G (K304E) mutation. The medication is sodium phenylbutyrate (ACER-001), which is currently FDA approved for the treatment of Urea Cyle Disorders. Previous research suggests that sodium phenylbutyrate may also be effective in the treatment MCADD. This study will investigate the safety and efficacy (how well it works) of sodium phenylbutyrate in patients with MCADD.

DETAILED DESCRIPTION:
Participation in the study will require three outpatient visits at the Clinical and Translational Research Center at the UPMC Children's Hospital of Pittsburgh (also called the PCTRC). The total length of the study participation is approximately 5 weeks.

Participants will come in for a screening visit (Visit 1) to where they will undergo some lab work testing to confirm they are eligible for the study. If it's determined that they are eligible, they will undergo training on the use of a continuous glucose monitor (CGM). They will be sent home and asked to wear the CGM for the next 10 days. This 10-day period is considered the run-in period.

Following the run-in period, participants will return to the site (Visit 2) in a fasting state. They will have an intravenous access line (IV) placed for several blood draws during the visit. Fasting labs will be drawn, then the participant will be provided with a meal and then will then be dosed with ACER-001. Following the dose of ACER-001, pharmacokinetics (PK) samples will be collected over the next 8 hours. Once the final PK sample has been collected, participant will be sent home with continuous glucose monitoring and will be asked to log their ACER-001 doses as well as overnight fasting times.

All participants will be dosed at 4.0 g/m2/day divided two times a day.

Participants will be asked to return approximately 2 weeks later for Visit 3 to complete the same procedures outlined for Visit 2.

Study staff will contact the participant by phone approximately 1 week after Visit 3 to follow up on any adverse events.

All study procedures will be done at no cost to the participants..

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of MCADD and molecular confirmation of at least one copy of the common c.985A>G mutation.
2. ≥4 years of age
3. Able to perform and comply with study activities placement of a continuous glucose monitor, IV catheter, and all blood draws.
4. Negative pregnancy test for all female subjects of childbearing age.
5. Signed informed consent by the subject or parent/guardian of minors.
6. All females of childbearing age and all sexually active males must agree to use an acceptable method of contraception throughout the study. Appropriate contraceptive methods include hormonal contraceptives (oral, injected, implanted, or transdermal), tubal ligation, intrauterine device, hysterectomy, vasectomy, or double barrier methods. Abstinence is an acceptable form of birth control, though appropriate contraception must be used if the subject becomes sexually active.
7. Willing and able to adhere to requirements for maintaining continuous glucose monitoring.

Exclusion Criteria:

1. Use of any investigational drug within 30 days of Day 1.
2. Active infection (viral or bacterial) or any other intercurrent condition as reported by the subject or noted on physical exam at screening.
3. Any clinical or laboratory abnormality of Grade 3 or greater severity according to the CTCAE v5.0, or Grade 3 elevations in liver enzymes, defined as levels 5-20 times ULN in alanine aminotransferase (ALT/SGPT), or aspartate aminotransferase (AST/SGOT) in a clinically stable subject.
4. Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at increased risk by participating in this study.
5. Use of any medication known to significantly affect renal clearance (e.g., probenecid) or to increase protein catabolism (e.g., corticosteroids), or other medication known to increase ammonia levels (e.g., valproic acid or haloperidol), within the 48 hours prior to Day 1 and throughout the study.
6. Subjects with renal insufficiency will be excluded from the study. Cutoff eGFR <60 mL/min/1.73m2 (GFR categories G3a-G5) will be used as measure of renal insufficiency.
7. Use of sodium benzoate within one week of Day 1.
8. Known hypersensitivity to PAA or PBA.
9. Breastfeeding or lactating females.
10. Subjects at risk of hypokalemia due to pre-existing diagnosis or on medications that can cause hypokalemia.
11. Subjects with type 1 or type 2 diabetes, or who take medications as part of their routine care that can cause hypoglycemia
12. A positive urine drug screen at screening for drugs without a prescription
13. Subjects who are taking medications in the antimetabolite drug class (e.g., hydroxyurea, 5-fluorouracil (5-FU), methotrexate) will be excluded; these medications can interfere with the DEXCOM sensor and cause inaccurate glucose readings

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE v5.0 | 5 weeks

SECONDARY OUTCOMES:
Length of time before glucose falls below 60 mg/dL | 5 weeks
  Comparison of the length of time each participant's glucose level stays above 60 mg/dL, comparing their values from the run-in period to the results obtained between Visits 2 and 3
Length of time before glucose falls below 70 mg/dL | 5 weeks
  Comparison of the length of time each participant's glucose level stays above 70 mg/dL, comparing their values from the run-in period to the results obtained between Visits 2 and 3
Length of time before glucose falls below 80 mg/dL | 5 weeks
  Comparison of the length of time each participant's glucose level stays above 80 mg/dL, comparing their values from the run-in period to the results obtained between Visits 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Vockley, MD, PhD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No